CLINICAL TRIAL: NCT05373914
Title: RESPIRARE - A Phase 2, Randomized, Double-blinded, Placebo-controlled, Efficacy and Safety Study of Cudetaxestat (BLD-0409) Assessed Across Three Dose Ranges With or Without Standard of Care (Nintedanib or Pirfenidone) in Patients With Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: RESPIRARE - Efficacy and Safety of Cudetaxestat in Patients With Idiopathic Pulmonary Fibrosis (IPF)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Blade Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B-0409-201
Record Dates: First submitted 2022-05-10; First posted 2022-05-13 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: IPF; Lung Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cudetaxestat (BLD-0409) 250mg once daily (Experimental): 250mg once daily (orally) with food
  Interventions: Drug: Cudetaxestat (BLD-0409); Drug: Control: Matching Placebo
- Cudetaxestat (BLD-0409) 500mg daily (Experimental): 500mg once daily (orally) with food
  Interventions: Drug: Cudetaxestat (BLD-0409); Drug: Control: Matching Placebo
- Cudetaxestat (BLD-0409) 500mg twice daily (Experimental): 500mg twice daily (orally) with food
  Interventions: Drug: Cudetaxestat (BLD-0409)
- Matching Placebo twice daily (Placebo Comparator): Matching placebo twice daily (orally) with food
  Interventions: Drug: Control: Matching Placebo

INTERVENTIONS:
Drug: Cudetaxestat (BLD-0409) — Cudetaxestat - 250mg tablets (orally)
  Other Names: Cudetaxestat
  Arms: Cudetaxestat (BLD-0409) 250mg once daily; Cudetaxestat (BLD-0409) 500mg daily; Cudetaxestat (BLD-0409) 500mg twice daily
Drug: Control: Matching Placebo — Placebo - 250mg tablets (orally)
  Arms: Cudetaxestat (BLD-0409) 250mg once daily; Cudetaxestat (BLD-0409) 500mg daily; Matching Placebo twice daily

SUMMARY:
The overall objective of this study is to evaluate the effectiveness and safety of cudetaxestat (BLD-0409) as compared to placebo with or without standard of care (nintedanib or pirfenidone) in subjects with idiopathic pulmonary fibrosis (IPF)

DETAILED DESCRIPTION:
This is a phase 2, randomized, double-blinded, placebo-controlled, efficacy and safety study of cudetaxestat (BLD-0409) assessed across three dose ranges with or without standard of care (nintedanib or pirfenidone) in patients with idiopathic pulmonary fibrosis (IPF). The study will include a screening period, a treatment period, and a follow-up period.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for participation in this study, subjects must meet all the following:

Age

1. At least 40 to 85 years of age, inclusive, at the time of signing the Informed Consent Form (ICF).

   Type of Subject and Disease Characteristics
2. Diagnosis of Idiopathic Pulmonary Fibrosis (IPF) as defined by ATS/ERS/JRS/ALAT guidelines.
3. IPF diagnosis within the past 7 years, with onset defined as the date of the first recorded diagnosis of IPF by HRCT and/or surgical biopsy or other appropriate tissue sample (e.g., cryobiopsy) in the medical history.
4. Interstitial pulmonary fibrosis defined by HRCT scan at Screening, with evidence of ≥10% to <50% parenchymal fibrosis (reticulation) and <25% honeycombing, within the whole lung. NOTE: HRCT scans will be assessed locally by the investigator prior to randomization. If a recent HRCT scan (within 3 months prior to Screening) is available, it can be utilized for screening purposes.
5. Observed time to disease progression (FVCpp) value >45% and <95% at Screening and Day 1 (prior to randomization).
6. Diffusing capacity of the lungs for carbon monoxide (DLCO) percent predicted and corrected by hemoglobin (Hb) value ≥25% and ≤90% at Screening (determined locally). If a DLCO is available within 3 months prior to Screening, it can be utilized for screening purposes. NOTE: Both FVC and DLCO testing must be representative of the IPF underlying disease (i.e., have been obtained in absence of an acute respiratory event [e.g., lung infection, cold]) or other events that are known to affect pulmonary function test (PFT) results (e.g., broken rib, chest pain, other).

   Contraception Related Contraception use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
7. Male subjects with partners of childbearing potential must use condom and female subjects of childbearing potential (including those <1 year postmenopausal) must use a highly effective method of contraception per Clinical Trial Facilitation Group (CTFG) recommendation during the conduct of the study, and for 30 days after the last dose of IP (males only during exposure to IP).

   Women not of childbearing potential are defined as:
   1. Post-menopausal women (defined as at least 12 months with no menses without an alternative medical cause); in women < 45 years of age, a high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy; OR
   2. Have had a hysterectomy and/or bilateral oophorectomy, bilateral salpingectomy, or bilateral tubal ligation/occlusion, at least 6 weeks prior to Screening; OR
   3. Have a congenital or acquired condition that prevents childbearing. Informed Consent
8. Capable of giving signed informed consent that includes compliance with the requirements and restrictions listed in the ICF and in this protocol Other
9. Treatment with approved background IPF therapy such as nintedanib or pirfenidone will be allowed as long as subjects are on a stable dose for at least 12 weeks prior to the first dose of the Investigational product and throughout the treatment period.

Exclusion Criteria:

Subjects meeting any of the following exclusion criteria are not eligible to be randomized into the study:

Medical Conditions

1. Evidence of significant obstructive lung disease by any of the following criteria: (1) forced expiratory volume in 1 second (FEV1)/FVC) ratio <0.70, or (2) extent of emphysema greater than the extent of fibrosis on HRCT. NOTE: This requires confirmation by the investigator prior to randomization.
2. Interstitial lung disease (ILD) other than IPF, including but not limited to any of the other types of idiopathic interstitial pneumonias; lung diseases related to exposure to fibrogenic agents or other environmental toxins or drugs; other types of occupational lung diseases; granulomatous lung diseases; pulmonary vascular diseases; systemic diseases, including vasculitis, infectious diseases, and connective tissue diseases. In cases of uncertain diagnosis, serological testing and/or review by multi-disciplinary team should be performed to confirm diagnosis of IPF vs. other types of ILD.
3. Sustained improvement in the severity of IPF during the 12 months prior to Screening, based on changes in FVC, DLCO, and/or HRCT scans of the chest.
4. History of other types of respiratory diseases, including diseases or disorders of the airways, lung parenchyma, pleural space, mediastinum, diaphragm, or chest wall that, in the opinion of the investigator, would impact the primary protocol endpoint or otherwise preclude the subject's participation in the study.
5. History of liver dysfunction including patients with moderate (Child Pugh B) or severe (Child Pugh C) impairment or disordered coagulation.
6. Medical conditions (e.g., myocardial infarction/stroke within the past 6 months), or logistical challenges that in the opinion of the investigator preclude the subject's adequate participation in the study.
7. Poorly controlled chronic heart failure (New York Heart Association Class 3 or above); clinical diagnosis of cor pulmonale requiring specific treatment; or severe pulmonary arterial hypertension requiring specific treatment that, in the opinion of the investigator, would preclude the subject's participation in the study.
8. Ongoing acute IPF exacerbation, or suspicion of such process during Screening or randomization, including hospitalization due to acute IPF exacerbation within 4 weeks prior to or during Screening.
9. High likelihood of lung transplantation (in the opinion of the Investigator) within 6 months after Day 1.
10. Body weight less than 40 kg (88.18 lb) or anorexia.
11. Any condition (other than IPF) that is likely to result in the death of the subject within the next year.
12. Any current malignancy (this does not include localized cancer such as basal or squamous cell carcinoma of skin). Any history of malignancy likely to result in mortality or requiring significant medical or surgical intervention within the next year.
13. The investigator judges that the subject will be unable to fully participate in the study and complete it for any reason, including inability to comply with study procedures and treatment, addiction, or any other relevant medical or psychiatric conditions.
14. Female subjects who are pregnant or breastfeeding.

    Diagnostic Assessments
15. The following laboratory parameters are excluded:

    1. Hb <10 g/dL (100 g/L)
    2. White blood cells (WBC) <3000/μL (<3000/mm3)
    3. Platelet count <70,000/μL (<70,000/mm3)
    4. Serum creatinine ≥1.5 x upper limit of normal (ULN)
    5. Glomerular filtration rate (GFR) < 60ml/m/1.73 or evidence of acute kidney injury
    6. Serum total bilirubin >1.5 x ULN
    7. Serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥2 x ULN, or serum alkaline phosphatase ≥2 x ULN.

    Excluded Therapies
16. Daily use of phosphodiesterase type 5 (PDE-5) inhibitor drugs (e.g., sildenafil, tadalafil) except for treatment of severe pulmonary artery hypertension
17. Use of any therapeutics with strong inhibitors and strong inducers of CYP3A4 or CYP2C8 [e.g., rifampicin, ketoconazole, phenytoin, ritonavir, macrolide antibiotics (e.g., telithromycin), and carbamazepine] is also prohibited.

    Prior/Concurrent Clinical Study Experience
18. Previous exposure to cudetaxestat
19. Use of any investigational drugs or unapproved therapies, or participation in a clinical study with an investigational new drug, within 30 days prior to first Screening visit.

    Other Exclusions
20. History of allergic or anaphylactic reaction to cudetaxestat, or to any component of the excipient.
21. History of intolerance to nintedanib or pirfenidone (e.g., arterial thromboembolic disease, bleeding, proteinuria, or photosensitivity)
22. Smoking within 3 months of Screening and/or unwilling to avoid smoking throughout the study

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-05-31 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Observed changes in FVC (L) from Baseline to Week 26 | Up to 182 days
  Change in Forced Vital Capacity FVC (L) from Baseline to Week 26.

SECONDARY OUTCOMES:
Observed time to disease progression (FVCpp) decline of ≥10% or death | Up to 182 days
  Time to disease progression
Observed time to disease progression (FVCpp) decline of ≥5% or death | Up to 182 days
  Time to disease progression.
Observed changes in Quantitative Lung Fibrosis (QLF) from Baseline to Week 26 | Up to 182 days
  Assessed by high-resolution computed tomography (HRCT)
Incidence, nature and severity of treatment-emergent adverse events (TEAEs) and Serious Adverse Events (SAEs) | Up to 182 days
  Safety and tolerability will be assessed based on the incidence, nature and severity of TEAEs and SAEs, and changes in safety laboratories, vitals and ECGs